CLINICAL TRIAL: NCT01339247
Title: Relative Bioavailability Study Between the Formulations: Paroxetine 25 mg Tablets With Controlled Release Manufactured by GSK Mississauga and Paroxetine 25 mg Tablets With Controlled Release Manufactured by SmithKline Beecham (Cidra), Fed Administration in Healthy Volunteers of Both Genders
Brief Title: Paxil CR Bioequivalence Study Brazil - Fed Administration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 114035
Record Dates: First submitted 2010-08-31; First posted 2011-04-20 (Estimated); Results first posted 2011-04-20 (Estimated); Last update posted 2018-06-20 (Actual); Status verified 2018-06

CONDITIONS: Depressive Disorder
Keywords: Bioequivalence; Paroxetine reference/test; healthy volunteers; Fed condition
MeSH Terms: conditions — Depressive Disorder | interventions — Paroxetine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Paxil CR Reference (Active Comparator): Paroxetine Hydrochloride 25 miligrams(mg) tablet with controlled release (Paxil CR), once a day, manufactured by SmithKline Beecham (Cork) Limited - Cidra - Puerto Rico, in Period 1, followed by Paroxetine Hydrochloride 25 mg tablet with controlled release (Paxil CR), once a day, manufactured by GlaxoSmithKline Inc. - Mississauga - Canada, in Period 2
  Interventions: Drug: Paxil CR 25 mg manufactured by SmithKline Beecham (Cork) Limited - Cidra - Puerto Rico; Drug: Paxil CR 25 mg manufactured by GlaxoSmithKline Inc. - Mississauga - Canada
- Paxil CR Test (Active Comparator): Paroxetine Hydrochloride 25 mg tablet with controlled release (Paxil CR), once a day, manufactured by GlaxoSmithKline Inc. - Mississauga - Canada, in Period 1, followed by Paroxetine Hydrochloride 25 miligrams(mg) tablet with controlled release (Paxil CR), once a day, manufactured by SmithKline Beecham (Cork) Limited - Cidra - Puerto Rico, in Period 2
  Interventions: Drug: Paxil CR 25 mg manufactured by SmithKline Beecham (Cork) Limited - Cidra - Puerto Rico; Drug: Paxil CR 25 mg manufactured by GlaxoSmithKline Inc. - Mississauga - Canada

INTERVENTIONS:
Drug: Paxil CR 25 mg manufactured by SmithKline Beecham (Cork) Limited - Cidra - Puerto Rico — Paroxetine Hydrochloride 25 miligrams(mg) tablet with controlled release (Paxil CR), once a day, manufactured by SmithKline Beecham (Cork) Limited - Cidra - Puerto Rico (reference formulation)
Drug: Paxil CR 25 mg manufactured by GlaxoSmithKline Inc. - Mississauga - Canada — Paroxetine Hydrochloride 25 mg tablet with controlled release (Paxil CR), once a day, manufactured by GlaxoSmithKline Inc. - Mississauga - Canada (test formulation)

SUMMARY:
The study is prospective, open, randomized, crossover in steady state and the volunteers received multiple doses of the test drug and the reference drug (two periods of drug administration after standardized meals).

DETAILED DESCRIPTION:
Title: Relative bioavailability study between the formulations: Paroxetine Hydrochloride 25 mg tablet with controlled release (Paxil CR) manufactured by GlaxoSmithKline Inc. - Mississauga - Canada (test formulation) and Paroxetine Hydrochloride 25 mg tablets with controlled release (Paxil CR) manufactured by SmithKline Beecham (Cork) Limited - Cidra - Puerto Rico (reference formulation), fed administration in healthy volunteers of both genders.

The study is prospective, open, randomized, crossover in steady state and the volunteers received multiple doses of the drug test and reference (two periods of drug administration). The population is composed of 60 healthy volunteers, adult of both gender, with age between 18 and 40 years, with a body mass index (BMI) between 18.5 and 27. Volunteers have weight above than 50 kg. 50% of the volunteers recruited are female and 50% male. There are no restrictions regarding the ethnic group.

The relative bioavailability of the formulations after oral administration in steady state will be evaluated based on statistical comparisons of relevant pharmacokinetic parameters obtained from data of drug concentration in blood. The concentration of Paroxetine hydrochloride (controlled release) will be measured by an appropriate analytical method and valid after the drug administration.The Pharmacokinetic samples will be collected at steady state in each period after standardized meals. The safety assessment will include evaluation and clinical monitoring, vital signs monitoring, ECG, and laboratory tests. Adverse events will be monitored throughout the study.

ELIGIBILITY:
EXCLUSION CRITERIA:

* hypersensitivity to the study drug or to compounds chemically related;
* history of serious adverse events;
* concurrent or recent use of other antidepressives, schizophrenia, anticonvulsant;
* History of liver, heart, gastrointestinal or renal illness;
* ECG findings not recommended according to the investigator judgement;
* The volunteer ingests more than 5 cups of coffee or tea a day.

INCLUSION CRITERIA:

* Man and woman (since they are not pregnant or breastfeeding);
* age between 18 and 40 years;
* non-smoker and not addict;
* mass index between 18,5 and 27;
* good health conditions or without significant illness, by judgement of a legally qualified professional;
* sign the informed consent.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2009-10-20 (Actual); Primary Completion 2009-11-16 (Actual); Study Completion 2009-11-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Belo Horizonte, Minas Gerais, Brazil

REFERENCES:
- See also: Results for study 114035 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/114035?search=study&search_terms=114035#rs

RESULTS

PARTICIPANT FLOW:
Groups:
- Test Product in Period 1; Reference Product in Period 2: Test product: paroxetine hydrochloride tablet with controlled release (Paxil CR) 25 milligrams (mg) manufactured by GlaxoSmithKline Inc. - Mississauga - Canada in Period 1; followed by reference product: Paxil CR 25 mg manufactured by SmithKline Beecham (Cork) Limited - Cidra - Puerto Rico in Period 2
- Reference Product in Period 1; Test Product in Period 2: Reference product: Paxil CR 25 mg manufactured by SmithKline Beecham (Cork) Limited - Cidra - Puerto Rico in Period 1; followed by test product: Paxil CR 25 mg manufactured by GlaxoSmithKline Inc. - Mississauga - Canada in Period 2
Period: Period 1
Arm/Group | Test Product in Period 1; Reference Product in Period 2 | Reference Product in Period 1; Test Product in Period 2
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Test Product in Period 1; Reference Product in Period 2 | Reference Product in Period 1; Test Product in Period 2
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Participants Receiving Both Test and Reference Product: Participants receiving either test product: Paxil CR 25 mg manufactured by GlaxoSmithKline Inc. - Mississauga - Canada in Period 1; followed by reference product: Paxil CR 25 mg manufactured by SmithKline Beecham (Cork) Limited - Cidra - Puerto Rico in Period 2 or reference product in Period 1 and test product in Period 2
Arm/Group | Participants Receiving Both Test and Reference Product
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: Years] | 27.73 (4.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 30
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 35
  Black | 4
  Mixed Race | 21

OUTCOME MEASURES:

1. Primary Outcome: AUC_ss
Description: The area under the plot of plasma concentration of drug against time after drug administration is defined as the area under the curve (AUC). The AUC_ss is the area under the curve during the steady-state period. The AUC_ss is of particular use in estimating the bioavailability of drugs, by measuring the extent of absorption. ng, nanograms; h, hour; ml, milliliter; ng.h/ml, nanograms per hour per milliliter.
Time Frame: Days 14 to 17 (period 1) and Days 23 to 24 (Period 2)
Population: Entire study population
Measure: Mean (Standard Deviation); unit: ng.h/ml
Groups:
- Test Product: Test product: Paxil CR 25 mg manufactured by GlaxoSmithKline Inc. - Mississauga - Canada in both periods
- Reference Product: Reference product: Paxil CR 25 mg manufactured by SmithKline Beecham (Cork) Limited - Cidra - Puerto Rico in both periods
Arm/Group | Test Product | Reference Product
Number analyzed (Participants) | 60 | 60
ng.h/ml | 672.9221 (432.2451) | 645.5407 (413.9084)
Statistical Analysis 1: Comparison: Test Product vs Reference Product; Test type: Non-Inferiority or Equivalence — This is a bioequivalence study. The study was performed to fulfill an official requirement of the Brazilian Regulatory Agency - ANVISA - upon a manufacturing site change; Ratio T formulation/R formulation = 1.0886, 90% CI 2-sided [1.0011 to 1.1770] — The ratio between the geometric means of the test (T) and reference (R) formulations was calculated

2. Primary Outcome: Cmin_ss
Description: Cmin_ss is defined as the minimum concentration of a drug observed after its administration, in steady-state. Cmin_ss is one of the parameters of particular use in estimating the bioavailability of drugs, for studies employing multiple doses.
Time Frame: Days 14 to 17 (period 1) and Days 23 to 24 (Period 2)
Population: Entire study population
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Test Product | Reference Product
Number analyzed (Participants) | 60 | 60
ng/ml | 19.4468 (13.7780) | 18.9010 (12.6797)
Statistical Analysis 1: Comparison: Test Product vs Reference Product; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio T formulation/R formulation = 1.0246, 90% CI 2-sided [0.9676 to 1.0849] — The ratio between the geometric means of the test (T) and reference (R) formulations was calculated

3. Primary Outcome: Cmax_ss
Description: Cmax_ss is defined as the maximum or "peak" concentration of a drug observed after its administration, in steady-state. Cmax_ss is one of the parameters of particular use in estimating the bioavailability of drugs, by measuring the total amount of drug absorbed.
Time Frame: Days 14 to 17 (period 1) and Days 23 to 24 (Period 2)
Population: Entire study population
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Test Product | Reference Product
Number analyzed (Participants) | 60 | 60
ng/ml | 36.7235 (21.0928) | 36.6630 (21.9946)
Statistical Analysis 1: Comparison: Test Product vs Reference Product; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio T formulation/R formulation = 1.0317, 90% CI 2-sided [0.9716 to 1.0956] — The ratio between the geometric means of the test (T) and reference (R) formulations was calculated

ADVERSE EVENTS:
Description: In order to simplify and avoid errors, the adverse events were separated by periods, not by sequences, due to the large number of adverse events.
Groups:
- Period 1: Participants receiving test product: Paxil CR 25 mg manufactured by GlaxoSmithKline Inc. - Mississauga - Canada or reference product: Paxil CR 25 mg manufactured by SmithKline Beecham (Cork) Limited - Cidra - Puerto Rico in Period 1
- Period 2: Participants receiving test product: Paxil CR 25 mg manufactured by GlaxoSmithKline Inc. - Mississauga - Canada or reference product: Paxil CR 25 mg manufactured by SmithKline Beecham (Cork) Limited - Cidra - Puerto Rico in Period 2
Arm/Group | Period 1 | Period 2
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 48/60 | 20/60
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Period 1 (N=60) | Period 2 (N=60)
Tachycardia (Cardiac disorders) | 0 | 1
Mydriasis (Eye disorders) | 1 | 0
Watery stools (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 16 | 0
Epigastralgia (Gastrointestinal disorders) | 4 | 0
Heartburn (Gastrointestinal disorders) | 3 | 0
Intestinal colic (Gastrointestinal disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Mild retch (Gastrointestinal disorders) | 1 | 0
Cephalea (General disorders) | 18 | 7
Fever (General disorders) | 1 | 0
Malaise (General disorders) | 3 | 0
Weakness (General disorders) | 0 | 1
Pain on the whole body (General disorders) | 0 | 1
Hyporexia (Metabolism and nutrition disorders) | 5 | 0
Lack of appetite (Metabolism and nutrition disorders) | 4 | 1
Somnolence (Nervous system disorders) | 22 | 8
Insomnia (Nervous system disorders) | 4 | 2
Dizziness (Nervous system disorders) | 0 | 3
Tremor (Nervous system disorders) | 2 | 1
Dysgeusia (Nervous system disorders) | 1 | 0
Thinking abnormal (Nervous system disorders) | 0 | 1
Sensation of slowness (Nervous system disorders) | 1 | 0
Irritability (Psychiatric disorders) | 1 | 0
Agitation (Psychiatric disorders) | 1 | 0
Menstrual colic (Reproductive system and breast disorders) | 1 | 0
Retardation of ejaculation (Reproductive system and breast disorders) | 1 | 0
Ejaculation difficulty (Reproductive system and breast disorders) | 2 | 1
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sore throat without evidence of infection (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sore throat with hyperaemia in tonsils (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Tonsillitis (Infections and infestations) | 2 | 0
Perspiration (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.